CLINICAL TRIAL: NCT04653272
Title: Simple Knee Value, a Simple Score for Functional Assessment of the Knee - Study SKV
Brief Title: Simple Knee Value, a Simple Score for Functional Assessment of the Knee
Acronym: SKV
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/19/0350
Record Dates: First submitted 2020-11-03; First posted 2020-12-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Knee Injuries
MeSH Terms: conditions — Knee Injuries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: * Patients aged 16 to 40 years with ACL anterior cruciate ligament rupture, meniscal injury, patella instability or dislocation (Young Adult group),
  * Patients over 55 years of age with gonarthrosis ("Senior" adults group).
  Interventions: Other: Questionnaire
- Control: * a group of "young" (16 to 40 years old)
  * "senior" (over 55 years old) adult controls
  * Everybody free of knee pathology.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients will be evaluated identically to routine care with reference tests (Lysholm-Tegner, and Knee injury and Osteoarthritis Outcome Score (KOSS) and, IKDC (Evaluation of knee ligament injuries). This is filled in without any external help. The questionnaire includes the Lysholm-Tegner (young adult group), IKDC and KOOS scores (young and senior adult groups).

SUMMARY:
The pre- and post-operative functional assessment of patients' knees is of great interest for the practitioner, whether it is in his or her daily practice to determine the appropriate management of the patient, or to conduct clinical studies. The scores used are established in several languages to provide a uniformly accepted unit of measurement.

DETAILED DESCRIPTION:
The pre- and post-operative functional assessment of patients' knees is of great interest for the practitioner, whether it is in his or her daily practice to determine the appropriate management of the patient, or to conduct clinical studies. The scores used are established in several languages to provide a uniformly accepted unit of measurement.

A large number of functional knee scores already exist. These include scores for Lysholm-Tegner, International Knee Documentation Committee (IKDC) and Knee injury and Osteoarthritis Outcome Score (KOOS), but these can be difficult to apply in practice. daily due to their length, which may be too time-consuming for the clinician when consultations for example.

Shoulder surgeons are familiar with the Simple Shoulder Value (SSV) score, which simply consists of asking the patient how much they value their shoulder on the day of the exam, compared to a normal shoulder in percentage terms. It has been shown to produce results that are close to Constant score or Rowe and American Shoulder Score and Elbow score Surgeons Score after shoulder surgery. It is, since its description, very much used in daily practice by shoulder surgeons because of its speed and simplicity of execution.

No such assessment exists to our knowledge for the knee. The validation of a score of this type for the knee joint would allow the use of a new practical tool for a better patient management while saving the practitioner and the patient money. time in consultation.

The investigators would like to propose a functional knee score similar to the ISS for the shoulder that would allow a self-assessment of the condition of a knee, compared to a normal knee in percentage terms.

The hypothesis is that the SKV (Simple Knee Value) is a valid score giving results of equivalent to the various scores already used in the functional assessment of the knee in the different pathological situations in adult and paediatric populations

ELIGIBILITY:
Inclusion Criteria:

For the patients:

1. Patients aged 16 to 40 years with ligament rupture anterior cruciate ACL, meniscal lesion, instability or anterior patella dislocation ("young" adult group),
2. Patients over 55 years of age with gonarthrosis. ("Senior" adults group).

For the controls:

In order to test the discriminating qualities of the SKV score, a group young" (16 to 40 years old) and "senior" (16 to 40 years old) adult witnesses, and 55 years old) with no problems with one of their knees.

For all participants :

* Understanding French
* Having given its non-opposition and for minors having obtained the non-opposition of one of the holders of parental authority
* Affiliation to a social security scheme

Exclusion Criteria:

For all participants :

* Memory disorders,
* Psychiatric disorders,
* Patient refusal to participate in the study,
* Patient under the protection of adults (guardianship, guardianship, safeguarding of justice),
* Pregnant and/or breastfeeding woman

Ages: 16 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 16 to 40 years with ligament rupture anterior cruciate ACL, meniscal lesion, instability or anterior patella dislocation ("young" adult group), and patients over 55 years of age with gonarthrosis. ("Senior" adults group).
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
SKV and score | Base line
  The analysis of the correlations between the SKV and the validated Functional Scores is based on the calculation of Spearman correlation coefficients.
SKV and score | 2 weeks
  The analysis of the correlations between the SKV and the validated Functional Scores is based on the calculation of Spearman correlation coefficients.
SKV and score | 2 months
  The analysis of the correlations between the SKV and the validated Functional Scores is based on the calculation of Spearman correlation coefficients.
SKV and score | 6 months
  The analysis of the correlations between the SKV and the validated Functional Scores is based on the calculation of Spearman correlation coefficients.

SECONDARY OUTCOMES:
SKV reproducibility | Base line
  The analysis of the reproducibility of the SKV score is based on the calculation of intraclass correlation coefficients in order to evaluate the concordance between the SKV score at inclusion and preoperatively in patients with a surgical indication.
SKV reproducibility | 6 months
  The analysis of the reproducibility of the SKV score is based on the calculation of intraclass correlation coefficients in order to evaluate the concordance between the SKV score at inclusion and preoperatively in patients with a surgical indication.
SKV sensitivity | Base line
  The analysis of the sensitivity to change in the SKV score is based on paired serial comparison tests (Wilcoxon test) of the SKV score at baseline and at 6 months postoperative follow-up in patients with a surgical indication.
SKV sensitivity | 6 months
  The analysis of the sensitivity to change in the SKV score is based on paired serial comparison tests (Wilcoxon test) of the SKV score at baseline and at 6 months postoperative follow-up in patients with a surgical indication.
SKV quality | base line
  The analysis of the discriminating qualities of the SKV score (and other functional scores) is based on a comparison of the distribution of the SKV score (and other functional scores) measured at inclusion in adult patients and adult controls.
SKV quality | 2 weeks
  The analysis of the discriminating qualities of the SKV score (and other functional scores) is based on a comparison of the distribution of the SKV score (and other functional scores) measured at inclusion in adult patients and adult controls.
SKV quality | 2 months
  The analysis of the discriminating qualities of the SKV score (and other functional scores) is based on a comparison of the distribution of the SKV score (and other functional scores) measured at inclusion in adult patients and adult controls.

CONTACTS AND LOCATIONS:
Overall Officials: Etienne CAVAIGNAC, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Etienne Cavaignac, Toulouse, France